CLINICAL TRIAL: NCT02304965
Title: Daily Physical Activity at Pulse Pressure Above an Individual Threshold in Patients With Continuous Flow Left Ventricular Assist Devices - a Feasibility Study
Brief Title: Activity at Pulse Pressure Above an Individual Threshold in Patients With LVAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU-B03
Record Dates: First submitted 2014-11-21; First posted 2014-12-02 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-06

CONDITIONS: Heart Failure
Keywords: LVAD
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Daily physical activity (Experimental): Eligible subjects will be included in the feasibility study to conduct an individualized and structured training program with defined walking and cycling on a bicycle ergometer for 2 months.
  Interventions: Behavioral: Daily physical activity

INTERVENTIONS:
Behavioral: Daily physical activity — A combination of walking (> 10.000 steps per day) and cycling on a stationary bicycle at home at an individual intensity. For the activity walking patients need to walk at a certain speed (e.g. 3 km/h) in order to be in the range of pulsatility as obtained from their pre-training treadmill test. For cycling a defined power in watt and duration will be given to each patient as defined from the pre-training cycling test.

SUMMARY:
Pilot study in patients with continuous flow left ventricular assist device (cfLVAD) to proof the feasibility of a specific individual training at home aimed to increase pulse pressure above a predefined threshold which might attenuate the loss of arterial wall thickness.

Hypothesis:

Increasing daily physical activity near to normal (> 10.000 steps per day) with a pre-defined level of pulse pressure (intensity) is a realizable and feasible approach to investigate changes in arterial wall thickness and cardio-respiratory capacity in cfLVAD patients.

DETAILED DESCRIPTION:
The investigators will study 3 cfLVAD patients with low pulse pressure during work package 1 using two different exercises, treadmill and bicycle. Walking and cycling present the most commonly used physical activities which are applicable to most individuals on a daily basis. The investigators aim to demonstrate that individual changes of pulse pressure during these types of exercise can be assessed in cfLVAD patients.

In a feasibility study (work package 2) the investigator will enroll 6 cfLVAD patients to perform home-based physical activity programs including walking a defined number of steps per day with a predefined speed and cycling with a predefined power [watt] on a bicycle ergometer. The performance of the patients will be monitored over seven days using a wearable activity device.

ELIGIBILITY:
Inclusion Criteria:

* age 45 to 65
* men
* time since cfLVAD implantation > 3 months and < 6 months
* low pulse pressure at rest, (no pulsatility)

Exclusion Criteria:

* musculoskeletal comorbidities restricting exercise
* known diabetes mellitus Type 1 and 2
* acute or chronic infections
* coronary heart disease before cfLVAD implantation
* no pulsatility with increasing exercise

Ages: 45 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-11; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in brachial artery smooth muscle thickness | At baseline and after 2 months
  Unit: mm

SECONDARY OUTCOMES:
Change from baseline in peak oxygen consumption | At baseline and after 2 months
  Unit: ml/min/kg
Change from baseline in pulse pressure during rest and exercise | At baseline and after 2 months
  Unit: mm/Hg
Change from baseline in daily physical activity | At baseline, after week 3, week 6, and after 2 months
  Unit: Steps per day assessed with a wearable activity device
Change from baseline in quality of life questionnaire (SF-36) | At baseline and after 2 months
  Unit: points

CONTACTS AND LOCATIONS:
Overall Officials: Sven Haufe, Dr., Principal Investigator — Hannover Medical School
Locations (1):
- Hannover Medical School, Hanover, Lower Saxony, Germany